CLINICAL TRIAL: NCT00425126
Title: Effect of Procrit(Epoetin Alfa) on Preventing Delayed Graft Function After Deceased Donor Renal Transplantation
Brief Title: Effect of Procrit (Epoetin Alfa) on Preventing Delayed Graft Function After Deceased Donor Renal Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: West Penn Allegheny Health System (Other)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: RC-4044
Record Dates: First submitted 2007-01-18; First posted 2007-01-22 (Estimated); Last update posted 2010-05-27 (Estimated); Status verified 2010-05

CONDITIONS: Delayed Graft Function
Keywords: Delayed Graft Function; Kidney Transplantation
MeSH Terms: conditions — Delayed Graft Function | interventions — Epoetin Alfa

INTERVENTIONS:
Drug: Epoetin Alfa

SUMMARY:
Delayed graft function (DGF) is a major complication following deceased donor renal transplantation. The surgical procedure of harvesting a kidney from a cadaveric donor and implanting the kidney into the recipient inevitably causes some amount of injury. While not always clinically significant, anywhere from 10-50% of transplant patients may develop DGF. Ongoing research in animal models has demonstrated benefit with administration of erythropoietin. The investigators propose to study the effect of Procrit(Epoetin Alfa) on delayed graft function in subjects undergoing kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting for kidney transplantation
* Age > 18
* Deceased donor kidney transplant

Exclusion Criteria:

* History of thrombosis or hypercoagulable state
* Receiving Coumadin or Heparin
* Hemoglobin >=14 g/dl
* Uncontrolled hypertension

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-02; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Decrease in Delayed Graft Function

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Marcus, MD, Principal Investigator — West Penn Allegheny Health System
Locations (1):
- Allegheny General Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] Sureshkumar KK, Hussain SM, Ko TY, Thai NL, Marcus RJ. Effect of high-dose erythropoietin on graft function after kidney transplantation: a randomized, double-blind clinical trial. Clin J Am Soc Nephrol. 2012 Sep;7(9):1498-506. doi: 10.2215/CJN.01360212. Epub 2012 Jun 28. PMID 22745272